CLINICAL TRIAL: NCT00732641
Title: Phase III Randomized, Prospective Multi-center Trial of PEG-Interferon α-2b as a Maintenance Therapy, Compared to Observation, in Patients With Multiple Myeloma Who Responded to Induction Therapy (Protocol No P01972)
Brief Title: Peginterferon α-2b as a Maintenance Therapy in Participants With Multiple Myeloma Who Responded to Induction Therapy (P01972-AM7)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01972
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Results first posted 2011-12-02 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peginterferon α-2b (Experimental): Peginterferon α-2b 35 μg, weekly, subcutaneous (SC), until disease progression or relapse, or for up to a maximum of 5 years.
  Interventions: Drug: Peginterferon
- No Treatment (No Intervention): Participants will be observed and will receive no treatment.

INTERVENTIONS:
Drug: Peginterferon — Peginterferon α-2b 35 μg, weekly, subcutaneous (SC), until disease progression or relapse, or for up to a maximum of 5 years.
  Arms: Peginterferon α-2b

SUMMARY:
This study aims to assess the efficacy of peginterferon α-2b, compared to a control arm not receiving any maintenance treatment, in adult subjects with multiple myeloma who have responded to a prior induction therapy. Peginterferon α-2b will be given once weekly as an injection until disease progression or relapse, or for up to a maximum of 5 years (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* Must demonstrate willingness to participate in the study and to adhere to dose and visit schedules
* Must be ≤85 years of age of either sex, and any race
* Must have stage II or III multiple myeloma with a histological confirmation consistent with the

diagnosis of multiple myeloma (by biopsy of an osteolytic or soft tissue tumour composed of plasma cells or bone marrow aspirate and/or biopsy demonstrating ≥ 10% plasmacytosis). The histological

confirmation should have been obtained prior to the induction chemotherapy or bone marrow transplant chemotherapy

* May not have received prior interferon for the treatment of multiple myeloma
* Must confirm that he/she is practicing adequate contraception
* If a female volunteer of childbearing potential, must have a negative serum pregnancy test

at Screening/Visit 1

-Must be free of any clinically relevant disease (other than multiple myeloma) that would, in the

principal investigator's and/or sponsor's opinion, interfere with the conduct of the study or study

evaluations

* Must be able to adhere to the dosing and visit schedules
* Clinical laboratory tests (complete blood chemistry [CBC], blood chemistries, urinalysis) must be

consistent with adequate hepatic and renal function, defined as <2 times upper limit of any laboratory normal (ULN) and adequate hematological functions defined as platelets > 50,000/mm^3, Hemoglobin ≥9.0 g/dL, white blood count (WBC) count ≥2000/mm^3

-Must have a complete, partial or minimal response after either one induction chemotherapy

regimen or one myelosuppressive chemotherapeutic treatment followed by peripheral blood stem cell

infusion as a first line treatment. Any type of pre-transplant chemotherapy and conditioning regimen is allowed

-Performance Status Karnofsky score of ≥60% at time of randomization

Exclusion Criteria:

* Is a female who is pregnant, or intends to become pregnant during the study
* Is nursing, or intends to be nursing during the study
* Has used any investigational product within 30 days prior to enrollment
* Have any of the following clinical conditions:

  * Pre existing psychiatric condition, especially depression, or a history of severe psychiatric disorder, such as major psychoses, suicidal ideation and/or suicidal attempt. Subjects with a history of mild depression may be considered for entry into the protocol provided that a pre-treatment assessment of the subject's mental status indicates that the subject is clinically stable and that there is ongoing evaluation of the patient's mental status during the study
  * Central Nervous System (CNS) trauma or active seizure disorders requiring medication
  * Significant cardiovascular dysfunction within the previous 6 months before the study starts (eg, angina, congestive heart failure, recent myocardial infarction, severe hypertension or significant arrhythmia) or patient with multigated acquisition (MUGA) or echocardiogram < 40%;
  * History of prior malignant disease within the previous 5 years before the study starts, except for surgically cured squamous cell or basal cell skin carcinoma or Stage I cervical carcinoma or cervical carcinoma in situ;
  * Known severe coagulation disorders, thrombophlebitis or pulmonary embolism or decompensate liver disease;
  * Uncontrolled diabetes mellitus or thyroid dysfunction (not responsive to therapy);
  * Severe chronic pulmonary disease (eg, chronic obstructive pulmonary disease);
  * Has active and/or uncontrolled infection
* Is in a situation or condition that, in the opinion of the investigator, may interfere with optimal

participation in the study

* Is participating in any other clinical study
* Is on the staff, affiliated with, or a family member of the staff personnel directly involved with this study
* Is allergic to or has sensitivity to the study drug or its excipients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2000-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- No Treatment: Participants were observed and received no treatment
Period: Overall Study
Arm/Group | Peginterferon α-2b | No Treatment
Started | 123 | 121
Completed | 17 | 9
Not Completed | 106 | 112
Not completed — Relapse or Progressive Disease | 65 | 101
Not completed — Serious Adverse Events | 12 | 3
Not completed — Physician Decision | 6 | 0
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Unable to Complete | 1 | 1
Not completed — Other | 18 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginterferon α-2b | No Treatment | Total
Number analyzed (Participants) | 122 | 121 | 243
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was for the intent-to-treat population (those who received at least one dose of study drug)
  years | 61.0 (8.5) | 62.3 (8.6) | 61.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender was for the intent-to-treat population (those who received at least one dose of study drug)
  Participants
    Female | 53 | 60 | 113
    Male | 69 | 61 | 130
Region of Enrollment [Number; unit: participants]
  Italy | 123 | 121 | 244

OUTCOME MEASURES:

1. Primary Outcome: Number of Days With Progression Free Survival (PFS)
Description: PFS was defined as response duration while on maintenance therapy. It was the length of time during and after treatment in which a participant was living with the cancer that did not get worse.
  PFS was calculated from the date of randomization to the date of the first documented tumor progression or relapse.
Time Frame: Baseline and up to 5 years (or to the date of the first documented tumor progression or relapse)
Population: Intent-to-treat population (those who received at least one dose of study drug)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Peginterferon α-2b | No Treatment
Number analyzed (Participants) | 122 | 121
Days | 1166 [682 to 1519] | 519 [403 to 634]

2. Secondary Outcome: Number of Days of Overall Survival (OS)
Description: OS was calculated from the date of randomization to the date of death for any
  cause. Participants alive at the end of study were censored at the last date they were known to be alive. Participants who were still living at the end of the study were censored on the last date they were known to be alive.
Time Frame: Baseline and up to 5 years (or to the date of the first documented tumor progression or relapse)
Population: Intent-to-treat population (those who received at least one dose of study drug)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Peginterferon α-2b | No Treatment
Number analyzed (Participants) | 122 | 121
Days | 2333 [2255 to NA] — not available - some participants were still living at the end of the study | 2329 [1539 to NA] — not available - some participants were still living at the end of the study

3. Secondary Outcome: Number of Participants With Complete Response (CR) to Treatment
Description: CR was defined as:
  * Absence of the original monoclonal paraprotein in serum and urine by immunofixation, maintained for a minimum of 6 weeks;
  * <5% plasma cells in a bone marrow aspirate and also on trephine bone biopsy, if biopsy was performed.
  * No increase in size or number of lytic bone lesions (development of a compression fracture did not include response);
  * Disappearance of soft tissue plasmocytomas.
Time Frame: Month 9 & Month 18
Population: Intent-to-treat population (those who received at least one dose of study drug)
Measure: Number; unit: Participants
Arm/Group | Peginterferon α-2b | No Treatment
Number analyzed (Participants) | 122 | 121
Participants
  Month 9 | 16 | 16
  Month 18 | 13 | 12

4. Secondary Outcome: Number of Participants With Partial Response (PR) to Treatment
Description: PR was defined as:
  * At least 50% reduction in the level of the serum monoclonal paraprotein, maintained for a minimum of 6 weeks;
  * Reduction in 24-hour urinary light chain excretion either by ≥ 90% or to < 200 mg, maintained for a minimum of 6 weeks;
  * For patients with non-secretory myeloma only, ≥ 50% reduction in plasma cells in a bone marrow aspirate and on a trephine biopsy, if biopsy was performed, maintained for a minimum of 6 weeks;
  * At least 50% reduction in the size of soft tissue plasmacytomas;
  * No increase in size or number of lytic bone lesions.
Time Frame: Month 9 & Month 18
Population: Intent-to-treat population (those who received at least one dose of study drug)
Measure: Number; unit: Participants
Arm/Group | Peginterferon α-2b | No Treatment
Number analyzed (Participants) | 122 | 121
Participants
  Month 9 | 65 | 54
  Month 18 | 45 | 29

5. Secondary Outcome: Number of Participants With Minimal Response (MR) to Treatment
Description: MR was defined as:
  * A 25-49% reduction in the level of the serum monoclonal paraprotein maintained for a minimum of 6 weeks;
  * Reduction in the 24-hour urinary light chain excretion, which still exceeded 200mg/24 hours, maintained for a minimum of 6 weeks;
  * For patients with non-secretory myeloma only, 25-49% reduction in plasma cells in a bone marrow aspirate and on a trephine biopsy, if biopsy was performed, maintained for a minimum of 6 weeks;
  * A 25-49% reduction in the size of soft tissue plasmacytomas;
  * No increase in the size or number of lityc lesions.
Time Frame: Month 9 & Month 18
Population: Intent-to-treat population (those who received at least one dose of study drug)
Measure: Number; unit: Participants
Arm/Group | Peginterferon α-2b | No Treatment
Number analyzed (Participants) | 122 | 121
Participants
  Month 9 | 5 | 4
  Month 18 | 1 | 3

6. Secondary Outcome: Number of Participants With Progressive Disease(PD) or Relapse From CR
Description: PD (for patients not in CR) required one or more of the following:
  * 25% increase in serum monoclonal paraprotein level, 24-hour urinary light chain excretion, or plasma cells;
  * Increase in size of existing or development of new bone lesions/soft tissue plasmacytomas;
  * Development of hypercalcemia.
  Relapse from CR required at least one of the following:
  * Reappearance of serum or urinary paraprotein;
  * >5% plasma cells;
  * Development of new lytic bone lesions or soft tissue plasmacytomas or increase in the size of residual bone lesions;
  * Development of hypercalcemia.
Time Frame: Month 9 & Month 18
Population: Intent-to-treat population (those who received at least one dose of study drug)
Measure: Number; unit: Participants
Arm/Group | Peginterferon α-2b | No Treatment
Number analyzed (Participants) | 122 | 121
Participants
  Month 9 | 36 | 47
  Month 18 | 63 | 77

7. Secondary Outcome: Quality of Life
Description: Participants were given the Europen Organization for Research in Cancer Therapy Quality of Life Questionnaire (EORTC QLQ), version 2.0, which consisted of 30 questions. The questionnaire evaluated global health/quality of life and incorporated five functional scales (Physical; Role; Emotional; Cognitive; Social). All of the scales ranged in score from 0 (worst) to 100 (best).
Time Frame: Screening and Last Observation (up to 5 years)
Population: Intent-to-treat population (those who received at least one dose of study drug).
  The number of participants analyzed varied depending on the number of observations available for each category.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Peginterferon α-2b | No Treatment
Number analyzed (Participants) | 122 | 121
Score on a scale
  Global Score (baseline) | 44.0 (12.5) | 45.2 (10.8)
  Global Score (last observation) | 41.4 (12.5) | 42.0 (10.6)
  Global Score (change) | -2.8 (15.5) | -2.6 (13.1)
  Physical Functioning Score (baseline) | 80.3 (22.9) | 74.0 (25.6)
  Physical Functioning Score (last observation) | 68.9 (29.0) | 68.7 (27.4)
  Physical Functioning Score (change) | -11.4 (28.5) | -6.9 (29.2)
  Role Functioning Score (baseline) | 85.4 (18.8) | 77.6 (25.0)
  Role Functioning Score (last observation) | 71.0 (30.1) | 72.2 (27.1)
  Role Functioning Score (change) | -14.1 (28.2) | -8.0 (31.0)
  Emotional Functioning Score (baseline) | 83.7 (15.9) | 80.9 (19.5)
  Emotional Functioning Score (last observation) | 72.6 (23.7) | 74.6 (20.7)
  Emotional Functioning Score (change) | -10.6 (19.1) | -8.0 (22.2)
  Cognitive Functioning Score (baseline) | 90.3 (14.9) | 89.3 (16.4)
  Cognitive Functioning Score (last observation) | 82.9 (20.9) | 84.2 (19.3)
  Cognitive Functioning Score (change) | -7.2 (17.8) | -7.5 (16.9)
  Social Functioning Score (baseline) | 86.0 (20.2) | 82.3 (24.0)
  Social Functioning Score (last observation) | 79.7 (25.9) | 82.6 (24.4)
  Social Functioning Score (change) | -6.4 (30.2) | -1.9 (27.6)

ADVERSE EVENTS:
Description: Tables contain both treatment-emergent events (events that occurred after receiving study drug) and non-treatment emergent events (events that occurred prior to receiving study drug).
Arm/Group | Peginterferon α-2b | No Treatment
Serious Adverse Events (participants affected / at risk) | 27/123 | 21/121
Other Adverse Events (participants affected / at risk) | 94/123 | 63/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon α-2b (N=123) | No Treatment (N=121)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
PRIMARY HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 1 (1) | 0 (0)
EYE PAIN (Eye disorders) | 1 (1) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 1 (1)
RETINAL VEIN THROMBOSIS (Eye disorders) | 1 (1) | 0 (0)
VISUAL ACUITY REDUCED (Eye disorders) | 0 (0) | 1 (1)
VISUAL IMPAIRMENT (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (2) | 0 (0)
CYST (General disorders) | 2 (2) | 0 (0)
DISEASE PROGRESSION (General disorders) | 4 (4) | 5 (5)
DISEASE RECURRENCE (General disorders) | 0 (0) | 1 (1)
INJECTION SITE NECROSIS (General disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 2 (2) | 1 (2)
SUDDEN CARDIAC DEATH (General disorders) | 0 (0) | 1 (1)
SWELLING (General disorders) | 0 (0) | 1 (1)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
LIVER DISORDER (Hepatobiliary disorders) | 0 (0) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 2 (2) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
HEPATITIS B (Infections and infestations) | 1 (1) | 1 (1)
HEPATITIS INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0)
MENINGITIS (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 0 (0) | 1 (1)
PSEUDOMONAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 (1) | 0 (0)
INTRAOCULAR PRESSURE INCREASED (Investigations) | 1 (1) | 0 (0)
CACHEXIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
GLIOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 1 (1)
PARKINSON'S DISEASE (Nervous system disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
THERAPEUTIC PROCEDURE (Surgical and medical procedures) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon α-2b (N=123) | No Treatment (N=121)
ANAEMIA (Blood and lymphatic system disorders) | 13 (13) | 15 (17)
LEUKOPENIA (Blood and lymphatic system disorders) | 9 (10) | 3 (3)
NEUTROPENIA (Blood and lymphatic system disorders) | 10 (12) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 15 (20) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 15 (20) | 3 (3)
ASTHENIA (General disorders) | 19 (26) | 3 (3)
FATIGUE (General disorders) | 8 (11) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 21 (36) | 9 (11)
PAIN (General disorders) | 7 (8) | 8 (8)
PYREXIA (General disorders) | 31 (51) | 19 (28)
HEPATOTOXICITY (Hepatobiliary disorders) | 7 (8) | 0 (0)
BRONCHITIS (Infections and infestations) | 11 (13) | 6 (12)
HERPES ZOSTER (Infections and infestations) | 6 (6) | 8 (9)
INFLUENZA (Infections and infestations) | 6 (7) | 10 (10)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 (11) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 13 (16) | 9 (14)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 7 (9)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 8 (8) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 8 (8) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator (PI) agrees not to publish/publicly present any interim study results without the sponsor's prior written consent. The PI further agrees to provide 45 days written notice to the sponsor prior to submission for publication/presentation to permit the sponsor to review copies of abstracts or manuscripts for publication which report any results of the Study. The sponsor shall have the right to review and comment on any presentation, which shall include editorial rights.